CLINICAL TRIAL: NCT06620081
Title: Effects of High-Flow Nasal Cannula on Exercise Outcomes in Lung Transplant Candidates: A Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital Israelita Albert Einstein (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 26495219.1.0000.0071
Record Dates: First submitted 2024-08-06; First posted 2024-10-01 (Actual); Last update posted 2024-10-01 (Actual); Status verified 2024-07

CONDITIONS: Pulmonary Diseases; Oxygen Therapy; High-flow Nasal Cannula; Exercise Tolerance
MeSH Terms: conditions — Lung Diseases

STUDY DESIGN:
Intervention Model Description: This pilot study is a randomized crossover clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Oxygen therapyHigh flow nasal cannula (Experimental): High-Flow Nasal Cannula Therapy (HFNC Therapy).
  Interventions: Other: Performance Tests; Other: Functional Tests
- Conventional oxygen therapy (Active Comparator): Conventional Oxygen Therapy with Venturi Mask or Non-Rebreather Mask.
  Interventions: Other: Performance Tests; Other: Functional Tests

INTERVENTIONS:
Other: Performance Tests — Three functional tests were performed: the six-minute walk test, incremental lower limb test with arterial blood gas analysis, and lower limb endurance test with inspiratory capacity measurement. Each test was conducted on different days with different devices: HFNC and conventional oxygen therapy, totaling six test days. The inspired oxygen fraction (FiO2) was titrated to maintain normoxia between 90% to 96% and was kept constant for both interfaces.
Other: Functional Tests — Three functional tests were performed: the six-minute walk test, incremental lower limb test with arterial blood gas analysis, and lower limb endurance test with inspiratory capacity measurement. Each test was conducted on different days with different devices: HFNC and conventional oxygen therapy, totaling six test days. The inspired oxygen fraction (FiO2) was titrated to maintain normoxia between 90% to 96% and was kept constant for both interfaces.

SUMMARY:
The study evaluated patients on the national lung transplant waiting list. It was pioneering in assessing high-complexity patients with severe pulmonary diseases subjected to a cardiopulmonary rehabilitation protocol using a treadmill. The main findings indicate that the distance covered in the six-minute walk test was greater when using the high-flow nasal cannula supplementation. The improvement in exercise performance in this group is associated with a reduction in arterial carbon dioxide, optimization of hydrogen potential, and a decrease in dynamic hyperinflation, leading to fewer symptoms of dyspnea.

DETAILED DESCRIPTION:
Introduction: Pulmonary diseases have a significant global prevalence, and lung transplantation is indicated for advanced cases. Rehabilitation is essential for patients on the waiting list and requires ventilatory devices for symptom control during exertion. The high-flow nasal cannula is a promising alternative, but its effects on exercise outcomes are uncertain. Objectives: To assess the effects of high-flow nasal cannula on the outcomes of the six-minute walk test. Method: A randomized crossover clinical trial evaluated ten volunteers listed on the national lung transplant waiting list. Three functional tests were performed: the six-minute walk test, incremental lower limb test with arterial blood gas analysis, and lower limb endurance test with inspiratory capacity measurement. Each test was conducted on different days with different devices: high-flow nasal cannula and conventional oxygen therapy, totaling six test days. The inspired oxygen fraction was titrated to maintain normoxia between 90% to 96% and was kept constant for both interfaces.

ELIGIBILITY:
Inclusion Criteria:

* Volunteers of both sexes
* Patients on the national lung transplant waiting list
* Chronic obstructive pulmonary disease
* Idiopathic or familial pulmonary fibrosis
* Bronchiectasis
* Sarcoidosis

Exclusion Criteria:

* Osteoarticular limitation,
* Neuromuscular disease,
* Anemia
* Hyperglycemia
* Arrhythmia
* Left heart failure
* Pulmonary hypertension

Ages: 30 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-06-02 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2024-07-24 (Actual)

PRIMARY OUTCOMES:
Evaluate the effect of HFNC on the distance covered in the 6MWT | 24 months
  Assessment of the distance traveled in 6 minutes.
Effect of HFNC on CO2 kinetics. | 24 months
  Assessment of the kinetics of effort-induced carbon dioxide.
Investigate the effect of HFNC on exercise-induced dynamic hyperinflation in patients on the lung transplant waiting list participating in a cardiopulmonary rehabilitation program. | 24 months
  Assessment of high-flow therapy in effort-induced hyperinflation.

CONTACTS AND LOCATIONS:
Overall Officials: Elaine Cristina Pereira, Study Chair — Albert Einstein Israelite Hospital; José Eduardo Afonso Júnior, Study Chair — Albert Einstein Israelite Hospital; Melline Della Torre de Almeida, Study Chair — Albert Einstein Israelite Hospital; Priscila Borelli Pereira Leite, Study Chair — Albert Einstein Israelite Hospital; Thaise de Lucca Cappeline, Study Chair — Albert Einstein Israelite Hospital; Thaís Melatto Loschi, Study Chair — Albert Einstein Israelite Hospital; Vanuza Ferreira dos Santos, Study Chair — Albert Einstein Israelite Hospital; Luciana Diniz Nagem Janot de Matos, Study Director — Albert Einstein Israelite Hospital
Locations (1):
- Albert Einstein Israelite Hospital, São Paulo, Brazil

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-06-19): https://cdn.clinicaltrials.gov/large-docs/81/NCT06620081/Prot_SAP_000.pdf
  • Informed Consent Form (2019-07-12): https://cdn.clinicaltrials.gov/large-docs/81/NCT06620081/ICF_001.pdf